CLINICAL TRIAL: NCT06210074
Title: Performance of Tampons as a Biospecimen Collection Tool for the Detection of Human Papillomavirus in a Colposcopy Setting
Acronym: PETAHG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampon Innovations Ltd (Industry)
Collaborators: University of Edinburgh (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Organization: Anne's Day Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PETAHG-ED-001
Record Dates: First submitted 2023-12-22; First posted 2024-01-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: CIN2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main Study Arm (Experimental): Women attending for routine colposcopy clinics as part of standard of care will be provided with the opportunity to participate and get tested with the Daye Diagnostic Tampon. Initial notice of the study will be via a patient information sheet sent with the colposcopy invitation
  Interventions: Device: Daye Diagnostic Tampon

INTERVENTIONS:
Device: Daye Diagnostic Tampon — The DAYE Diagnostic Tampon is a class A in vitro diagnostic device. It has CE certification (self-certified via a declaration of conformity, following the IVDR (EU) 2017/746).
  The DDT is constructed entirely from woven cotton and consists of an absorbent core wrapped in a protective sleeve. The DDT is loaded in an applicator to aid with insertion. The DDT needs to be worn for 20 minutes then when removed should be placed immediately in the sterile container.

SUMMARY:
Evaluation of the clinical performance of the Daye Diagnostic Tampon (DDT) for the detection of Human Papilloma Virus (HPV) infection associated with high grade cervical disease. Cross sectional design with comparison to a clinician taken biospecimen. Performance will be measured relative to the presence/absence of histologically confirmed disease

DETAILED DESCRIPTION:
Type of Study: Clinical Trial

Goal: The goal of this clinical trial is to evaluate the clinical performance of the Daye Diagnostic Tampon (DDT) for the detection of HPV infection associated with high-grade cervical disease.

Main Questions:

What is the sensitivity and specificity of molecular HPV assays in detecting high-grade cervical disease (CIN2+) using the DDT compared to a clinician-taken, liquid-based cytology (LBC) sample?

How does the relative sensitivity and specificity of HPV detection in the tampon compare to the LBC sample for the detection of CIN2+?

Participants:

Women attending routine colposcopy clinics as part of standard care.

Main Tasks:

Provide informed consent. Undergo routine colposcopy. Use the DAYE Diagnostic Tampon (DDT). Provide a clinician-taken liquid-based cytology (LBC) sample. Complete a short questionnaire.

Comparison Group:

Researchers will compare the performance of the DAYE Diagnostic Tampon (DDT) to a clinician-taken, liquid-based cytology (LBC) sample to determine if there are differences in sensitivity and specificity for the detection of high-grade cervical disease (CIN2+). The comparison will assess the relative sensitivity and specificity of HPV detection in the tampon versus the LBC sample for the presence/absence of histologically confirmed disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 25-65 years (inclusive)
* Ability to understand patient information sheet
* Ability to provide informed consent
* Natal female
* Referred to colposcopy for routine indications
* In-tact cervix

Exclusion Criteria:

* <25 years of age or over 65 years of age
* Hysterectomised
* Known allergy or sensitivity to tampons
* Pregnancy (current) or within last 3 months
* History of toxic shock syndrome
* Concurrent participation in other interventional research project

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals aged 25-65 years (inclusive Ability to understand patient information sheet Ability to provide informed consent Natal female Referred to colposcopy for routine indications In-tact cervix
Enrollment: 250 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity (%) of the tampon-assay combination & LBC assay combination for detection of histologically high grade disease | end of study (12 months from start)
  To assess the sensitivity and specificity of molecular HPV assays for the detection of high grade cervical disease (defined as cervical intraepithelial neoplasia grade 2 or worse, CIN2+) using the DDT AND a clinician taken, liquid based cytology (LBC) sample
Relative sensitivity of the tampon-assay combination vs the LBC-assay combination | end of study (12 months from start)
  To determine the relative sensitivity and specificity of HPV detection in the tampon vs the LBC sample for the detection of CIN2+.

SECONDARY OUTCOMES:
Attitudes to using the Diagnostic Tampon | up to 24 weeks
  Reponses/scores derived from brief questionnaire to assess the attitudes of the study recruits to the use of the DDT for HPV sampling
Assessment of Participation Willingness in Research on Tampon-Based Microbial Testing Among Colposcopy Patients | up to 24 weeks
  Quantification of Participation Rates: A comparison between the number of colposcopy patients invited to participate and those who actively engaged in research. This study aims to determine the level of willingness within the colposcopy population to partake in research focused on the utilization of tampons for microbial testing. The outcome measure will specifically assess the percentage of invited participants who actively contribute to the study, shedding light on the feasibility and acceptance of the proposed research intervention within this demographic. This quantification will be instrumental in understanding the potential for successful recruitment and engagement in future studies involving tampon-based microbial testing.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Cuscieri, Principal Investigator — NHS Lothian

IPD SHARING:
Plan to Share IPD: Undecided